CLINICAL TRIAL: NCT02182986
Title: Biomarkers for Post-Transplant Lymphoproliferative Disorders in Children (CTOTC-06)
Brief Title: Biomarkers for Post-Transplant Lymphoproliferative Disorders in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-06
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Heart Transplant; Small Intestine Transplant; Kidney Transplant; Liver Transplant; EBV-Related PTLD; PTLDs
Keywords: Biomarkers; Post-Transplant Lymphoproliferative Disorders (PTLDs)
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects Enrolled Pre-Transplant: Subjects (N=approximately 357) Enrolled Pre-Transplant
  * Subjects with evidence of EBV infection prior to transplant
  * Subjects without evidence of EBV infection prior to transplant, who are at risk of developing EBV infection after transplant
  Interventions: Procedure: transplant; Drug: Immunosuppressive Drugs
- Subjects Enrolled Post-Transplant: Subjects (N=approximately 588) Enrolled 3 Yrs Post-Transplant
  * Subjects with evidence of EBV infection prior to transplant
  * Subjects without evidence of EBV infection prior to transplant, who are at risk of developing EBV infection after transplant
  Interventions: Procedure: transplant; Drug: Immunosuppressive Drugs

INTERVENTIONS:
Procedure: transplant — All subjects enrolled in this study are candidates for/recipients of solid organ transplants as a therapeutic for end stage diseases (e.g., heart, liver, heart with liver, kidney, small intestine, or liver with small intestine transplants).
  Other Names: transplantation
Drug: Immunosuppressive Drugs — Immunosuppressive drugs prescribed as standard of care to prevent rejection of the allograft.
  Other Names: Immunosuppressive Medications

SUMMARY:
Solid organ transplantation is an important therapeutic option for children with a variety of end stage diseases. However, the same immunosuppressive medications that are required to prevent the child's immune system from attacking and rejecting the transplanted organ can predispose these individuals to developing a very serious cancer that is linked to Epstein-Barr virus (EBV).

DETAILED DESCRIPTION:
EBV-associated post-transplant lymphoproliferative disease (PTLD) is the most common malignancy in children after transplant. Diagnosis and effective treatment of the EBV-associated cancer is hampered by our inability to determine which children are at risk of developing these cancers and to detect the cancer at an early stage. In this study, we plan to test new "biomarkers" in the blood of children that will tell us very early on if the child is at risk of developing the EBV-associated cancer or if the cancer is present. These studies provide new opportunities for detection, diagnosis, and treatment of children with EBV-associated, post-transplant cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent or legal guardian must be able to understand and provide informed consent/assent;
* Candidate for or recipient of: heart, liver, heart with liver, small intestine, liver with small intestine, or kidney; and
* Subject enrolled within 3 years of transplant.

Exclusion Criteria:

* Previous diagnosis of PTLD;
* Transplant recipients of lung alone, or in combination with an eligible organ type;
* Pancreas transplantation with the exception of 'en bloc' transplant in combined liver and small intestine multivisceral transplantation;
* Any combination other than listed in inclusion criteria;
* History of any previous solid organ, stem cell, or bone marrow transplantation;
* Inability or unwillingness of the legal guardian and/or the subject to comply with the study protocol.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Candidates for or recipients of heart, liver, heart with liver, kidney, small intestine, or liver with small intestine at participating major pediatric solid organ transplant programs
Sampling Method: Non-Probability Sample
Enrollment: 944 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Epstein-Barr Virus (EBV) Positive Post-Transplant Lymphoproliferative Disorders (PTLD) | Receipt of transplanted organ(s) to confirmation of EBV-positive PTLD, up to year 4 post - enrollment
  The development of EBV positive PTLD during the study period as assessed by the local site pathologist, with confirmation of the PTLD diagnosis by the Study Clinicopathological Review Board (SCPRB)
Specified Gain-of-Function Mutations in EBV Latent Membrane Protein 1 (LMP-1) | Receipt of transplanted organ(s) to confirmation of mutations in EBV LMP1 , up to year 4 post - enrollment
  Specified gain-of-function mutations in EBV LMP-1 (e.g., corresponding to EBV LMP-1 variants G212S or S366T) detected by polymerase chain reaction (PCR) method
Pathogenic Changes in B Cell Clonotype Development | Receipt of transplanted organ(s) to confirmation of changes in B cell clonotype development, up to year 4 post - enrollment
  Pathogenic changes in B cell clonotype development as assessed using high throughput sequencing (HTS)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Esquivel, M.D., Ph.D., Principal Investigator — Stanford University; Daniel Bernstein, M.D., Study Chair — Stanford University
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford, Stanford, California
  - Medstar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - University of Miami Health System, Miami, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Derived] Rao M, Amouzgar M, Harden JT, Lapasaran MG, Trickey A, Armstrong B, Odim J, Debnam T, Esquivel CO, Bendall SC, Martinez OM, Krams SM. High-dimensional profiling of pediatric immune responses to solid organ transplantation. Cell Rep Med. 2023 Aug 15;4(8):101147. doi: 10.1016/j.xcrm.2023.101147. Epub 2023 Aug 7. PMID 37552988
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) — http://www.ctotc.org/